CLINICAL TRIAL: NCT00449098
Title: Comparative Study of the Safety and Effectiveness Between Ologen (OculusGen) Collagen Matrix Implant and Mitomycin-C in Glaucoma Filtering Surgery
Brief Title: Ologen (OculusGen)-Glaucoma MMC Control Trial in India
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mediking 0701; OculusGen-2006-02-20
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Collagen matrix; ologen; OculusGen; Trabeculectomy; anti scarring; tissue engineering; high risk patient for trabeculectomy; Aeon Astron
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

ARMS (2):
- OculusGen Biodegradable Collagen Matrix Implant (Experimental): Trabeculectomy with OculusGen Biodegradable Collagen Matrix Implant
  Interventions: Device: OculusGen Biodegradable Collagen Matrix Implant
- MMC (Active Comparator): Trabeculectomy with MMC
  Interventions: Drug: Trabeculectomy with MMC

INTERVENTIONS:
Device: OculusGen Biodegradable Collagen Matrix Implant — Trabeculectomy with OculusGen Biodegradable Collagen Matrix Implant
  Arms: OculusGen Biodegradable Collagen Matrix Implant
Drug: Trabeculectomy with MMC — Trabeculectomy with MMC
  Arms: MMC

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the ologen (OculusGen) Biodegradable Collagen Matrix Implant and the MMC group in filtration surgery.

DETAILED DESCRIPTION:
1. Study Objective: To compare the safety and effectiveness of the ologen (OculusGen) Biodegradable Collagen Matrix Implant and the MMC group in filtration surgery. The primary endpoint is to prove the effectiveness via the reduction of IOP, and the secondary endpoint is to prove the safety via the incidence of complications and adverse events.
2. Study Design: The study is designed as an open-label, randomized, parallel, comparative study. Patients who meet the inclusion/exclusion criteria and sign informed consent will be included. After enrollment, patients will be randomized into two groups: trabeculectomy with ologen (OculusGen) implant or trabeculectomy with mitomycin-C.
3. Follow-Up: There will be 7 post-operative and follow-up visits within 6 months of surgery: postoperative days 1, 7, 14, 30, 60, 90 and 180. A window of ± 7 days is allowed for the 30, 60, 90 day visits and ± 14 days for the 180 day visits. Further follow-up of subjects after the trial will be the responsibility of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over.
* Uncontrolled glaucoma, with failed medical and laser treatment, requiring trabeculectomy.
* Subject able and willing to cooperate with investigation plan.
* Subject able and willing to complete postoperative follow-up requirements.
* Subject willing to sign informed consent form.

Exclusion Criteria:

* Known allergic reaction to mitomycin-C or porcine collagen.
* Subject is on warfarin and discontinuation is not recommended.
* Normal tension glaucoma.
* Participation in an investigational study during the 30 days preceding trabeculectomy.
* Ocular infection within 14 days prior to trabeculectomy.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
the effectiveness via the reduction of IOP | 180 day

SECONDARY OUTCOMES:
the safety via the incidence of complications and adverse events. | 180 day

CONTACTS AND LOCATIONS:
Overall Officials: Rajul S Parikh, MD, Principal Investigator — V. S. T. Glaucoma Services, L. V. Prasad Eye Institute,
Locations (1):
- L. V. Prasad Eye Institute, Hyderabad, Andhra Pradesh, India

REFERENCES:
- [Result] Chen HS, Ritch R, Krupin T, Hsu WC. Control of filtering bleb structure through tissue bioengineering: An animal model. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5310-4. doi: 10.1167/iovs.06-0378. PMID 17122118
- [Result] Hsu WC, Spilker MH, Yannas IV, Rubin PA. Inhibition of conjunctival scarring and contraction by a porous collagen-glycosaminoglycan implant. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2404-11. PMID 10937547
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740